CLINICAL TRIAL: NCT06923072
Title: A Phase IIa Trial of Baricitinib in the Treatment of Kohlmeier-Degos Disease Patients With Neurological Involvement
Brief Title: Baricitinib in the Treatment of Kohlmeier-Degos Disease in Patients With Neurological Involvement
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002416; 002416-H
Record Dates: First submitted 2025-04-10; First posted 2025-04-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-19

CONDITIONS: Kohlmeier-Degos Disease; Malignant Atrophic Papulosis; Degos Disease; Papulosis, Malignant Atrophic
Keywords: Degos Disease; Kohlmeier-Degos; Baricitinib; Neurological involvement of Degos Disease
MeSH Terms: conditions — Malignant Atrophic Papulosis | interventions — baricitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with K(SqrRoot)(Delta)hlmeier-Degos Disease receiving Baricitinib (Experimental): All participants will take baricitinib 4mg oral daily for 24 weeks.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Participants will be instructed to take baricitinib 4mg oral daily for 24 weeks (with or without food)

SUMMARY:
Background:

Kohlmeier-Degos (KD) is a rare disease that causes inflammation and blood clots, leading to blockages in small blood vessels. These blockages can result in K-D lesions throughout the body, affecting the skin, lungs, heart, spinal cord, and brain. KD can be fatal. No treatment exists for this disease.

Objective:

To test a study drug (baricitinib) in people with brain and spine lesions caused by KD disease. Baricitinib is FDA approved to treat other disorders but has not yet been tried in people with KD.

Eligibility:

People aged 18 years or older with KD-related lesions in the brain and spine.

Design:

Participants will be screened; they will have a physical exam with blood tests. They will also have a baseline visit that may include multiple tests, such as imaging scans of the brain and spine; a lumbar puncture to collect fluid from the spinal canal; and a meeting with a neurologist. They will fill out a questionnaire about their health. They will continue to take their normal medications throughout the study.

Baricitinib is a tablet taken by mouth. Participants will remain on their normal medications for 12 weeks after their baseline visit. Then they will also take the study drug once a day at home for 24 weeks.

Participants will have clinic visits every few weeks for up to 40 weeks. Some visits may take 1 to 4 days. Baseline tests will be repeated 3 more times during study visits. Other visits will require only blood tests; these may be done by local labs that will send the samples to NIH; 2 visits may be done via telehealth....

DETAILED DESCRIPTION:
Study Description:

This phase II study will provide off-label baricitinib treatment in patients with Kohlmeier Degos disease (K-D) with neurologic involvement. We will perform a baseline research evaluation at the time of enrollment and follow each patient for 12 weeks of background therapy (defined as medications taken by the subject for management of Degos symptoms) followed by 24 weeks of baricitinib treatment (4 mg daily) in addition to background therapy followed by 4 additional weeks of background therapy with final safety assessment at 40 weeks. We will repeat research evaluations at the end of weeks 12, 24, and 36. We will compare the disease progression between weeks 1 through 12 to weeks 13 through 24 as well as weeks 13 through 36. We hypothesize that baricitinib, which targets type I interferon (IFN) and IFN-g signaling, will attenuate various neurological manifestations of K-D that are observed clinically, radiologically or in abnormal laboratory findings in our KD patients. This will help reduce IFN signaling in a manner that may slow or halt the disease progression as measured by the endpoints established below.

Objectives:

Primary Objective:

To test whether baricitinib delays progression of neuroradiological manifestations in patients with neurological involvement of K-D disease.

Secondary Objectives:

To test whether baricitinib treatment improves patient-reported outcomes.

Exploratory Objectives:

* Assess changes in immune cell proportion using single cell Ribonucleic Acid (RNA) sequencing (scRNA-seq) in biospecimens such as skin, cerebrospinal fluid (CSF) and blood after 12 and 24 weeks of baricitinib treatment compared to 12 weeks of just background therapy
* Assess changes in plasma/serum cytokine levels and IFN scores as well as biomarker assays in CSF/blood samples after 12 and 24 weeks of baricitinib treatment compared to 12 weeks of just background therapy.
* To assess whether 12 or 24 weeks of baricitinib treatment will stabilize or improve clinical neurologic exams.
* To assess whether 12 or 24 weeks of baricitinib treatment compared to 12 weeks of just background therapy will reduce the number of new acute K-D skin lesions or slow/halt the progression of existing K-D skin lesions. To assess whether 12 or 24 weeks of baricitinib treatment will reduce the number of new acute K-D skin lesions or slow/halt the progression of existing K-D skin lesions.

Endpoints:

* The primary endpoint will assess the stability of existing enhancing lesions or the lack of development of new enhancing lesions in the brain and spine observed by Magnetic Resonance Imaging (MRI) after 12 or 24 weeks of baricitinib treatment (4 milligrams [mg] daily) compared to existing enhancing lesions observed over 12 weeks of background therapy.
* The secondary endpoints will assess the change over 12 and 24 weeks of baricitinib treatment as compared to 12 weeks of background therapy only for the following outcomes: self-reported outcome measures based on health-related questionnaire ( SF-36 ).
* Exploratory endpoints of this study will be clinical and potential surrogate biomarker efficacy data, including:

  * Changes in transcriptome/ribonucleic acid (RNA) expression determined by scRNA-seq in skin, CSF and peripheral blood mononuclear cells (PBMCs) after 12 or 24 weeks of baricitinib treatment as compared to 12 weeks of background therapy only.
  * Attenuation of plasma/serum cytokine levels and IFN scores as well as biomarkers in assays using CSF and blood samples after 12 and 24 weeks of baricitinib treatment as compared to 12 weeks of background therapy.
  * Stability or improvement of motor and/or sensory function on clinical neurologic exams after the 12 or 24 weeks of baricitinib treatment as compared to 12 weeks of background therapy only.
  * Changes in the number of new acute K-D skin lesions or slowing/halting progression of existing K-D skin lesions after 12 or 24 weeks of baricitinib treatment as compared to 12 weeks of background therapy only.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form by the subject or Legally Authorized Representative (LAR).
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 18 or older.
* Subjects diagnosed with systemic Degos disease, who manifest neurologic abnormalities observed clinically, radiologically or in abnormal laboratory findings.
* Ability to take oral medication and be willing to adhere to the baricitinib regimen.
* For female patients of reproductive potential, non-pregnant, non-breastfeeding: agree to use of highly effective contraception for the duration of the study and 30 days after the last dose.
* Ability of subject or LAR to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Active infection not responding to appropriate therapy
* Hemoglobin <7 g/dL
* Platelet counts < 50 K /mcL
* Neutropenia (ANC <0.5 x k/mcL)
* Lymphopenia (Absolute Lymphocyte Count [ALC] <0.2x k/mcL)
* Liver function tests (LFTs > 2x time upper limit of normal)
* Estimated Glomerular Filtration Rate (eGFR)/Creatinine (Cr < 30 mL/min)
* Have experienced any of the following within 12 weeks of screening: VTE (DVT/pulmonary embolism [PE]), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have had symptomatic herpes zoster infection within 12 weeks prior to a enrolling in the study .
* Have had household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB.
* Have evidence of active TB or latent TB
* Have been exposed to a live vaccine within 12 weeks of baricitinib treatment or are expected to need/receive a live vaccine during the course of the study
* No gadolinium based contrast agent exposure is permitted if eGFR < 30 mL/min/1.73m^2 using the CKD-EPI equation measured within 5 days .
* Breast feeding
* Pregnancy
* Uncontrolled malignancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-12-14 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with stability of existing enhancing lesions in the brain and/or spine observed in MRI | Baseline, Week 12, Week 24, Week 36
  Stability of existing enhancing lesions in the brain and/or spine observed in MRI after 12 or 24 weeks of baricitinib treatment (4 mg daily) as compared to MRI images after 12 weeks of background therapy only.
Number of participants with no new enhancing lesions in the brain and/or spine observed in MRI | Baseline, Week 12, Week 24, Week 36
  Lack of development of new enhancing lesions in the brain and/or spine observed in MRI after 12 or 24 weeks of baricitinib treatment (4 mg daily) as compared to MRI images after 12 weeks of background therapy only.

SECONDARY OUTCOMES:
Change in health outcome questionnaire, Short Form-36 (SF-36) | Baseline, Week 12, Week 16, Week 24, Week 36, and up to Week 40
  Compare the change in health outcome questionnaire, Short Form-36 (SF-36), over 12 and 24 weeks of baricitinib treatment as compared to 12 weeks of background therapy. This 36-item, patient-reported survey assesses quality of life. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Neurological symptoms using CTCAE | Up to 40 weeks
  Compare the change of neurological symptoms using CTCAE over 12 and 24 weeks of baricitinib treatment as compared to 12 weeks of background therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia D Cudrici, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting approximately 6 months after publication and available indefinitely
Access Criteria: Data will be shared through the NHLBI BioData Catalyst, which is a controlled access repository.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002416-H.html